CLINICAL TRIAL: NCT04710459
Title: The Value of Endobronchial Cryotherapy in the Management of Malignant Endobronchial Obstruction in Patients With Inoperable NSCLC: A Prospective Analysis of Clinical and Survival Outcomes
Brief Title: Endobronchial Cryotherapy in Management of MEBO in Patients With Inoperable NSCLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Abdel Bary Ahmed Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abdel Bary Ahmed Ibrahim, Associate professor, South Valley University
Organization: South Valley University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVU-MED-84-10-12-2016
Record Dates: First submitted 2020-04-16; First posted 2021-01-14 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Non Small Cell Lung Cancer; Non-Small Cell Carcinoma of Lung, TNM Stage 4; Bronchogenic Cancer
Keywords: Non-small cell lung cancer (NSCLC); Cryotherapy; Chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): it included 30 patients, they were subjected to chemoradiotherapy plus endobronchial cryotherapy.
  Interventions: Procedure: cryotherapy
- Group 2 (No Intervention): it included include 30 patients, they were subjected to chemoradiotherapy.

INTERVENTIONS:
Procedure: cryotherapy — Group 1 included 30 patients, they were subjected to chemoradiotherapy plus endobronchial cryotherapy. Group 2 included include 30 patients, they were subjected to chemoradiotherapy.
  Arms: Group 1

SUMMARY:
Background: In end-stage patients when all management options have been used, will often develop compromise of their airways as the cancer continues to progress. Endobronchial therapy options may help to relieve some of their symptoms, allowing improvement in their shortness of breath as they go home in combination with other palliative therapies.

Objective: to compare the safety ; efficacy; and clinical outcome of endobronchial cryotherapy combined with chemotherapy and/ or radiotherapy versus chemo-radiotherapy alone on patients with Non small cell lung cancer.

Patients and method(s): A prospective randomized clinical trial was carried out on 60 patients with different ages of both sexes, diagnosed as bronchogenic carcinoma non-small cell lung cancer type (NSCLC) . The patients attended the hospital in the chest department, Qena Faculty of Medicine, South Valley University. Assessment of the patients was done and randomly assigned into two groups. Group1 ,Include 30 patients subjected to chemotherapy , radiotherapy and endobronchial cryotherapy.Group 2 , Include include 30 patients subjected to chemotherapy and radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* All cases with pathologically proved and inoperable NSCLC cases based on tumor position; in the main and subsegmental bronchi.

Exclusion Criteria:

* Cases with severe respiratory distress, uncorrectable impaired bleeding profile and prechemotherapy.

Ages: 47 Years to 71 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical changes of the cases after procedure. | the symptoms were evaluated before therapy as a baseline; and evaluated 4 weeks after procedure.
  Evaluation of the rate of symptoms relief after therapy
Respiratory function test evaluation | Change from Baseline Spirometry done before management, was compared with that was done at 4 weeks after management.
  Spirometry was done (FEV1 in %, FVC in %, FEV1/FVC in %).
Assessment of the overall survival | The overall survival was measured by the percentage of patients who still alive for 12 months after they were started the management.
  Assessment of the overall survival was done by Kaplan-Meier method
Assessment of the performance status | The mean Karnofsky performance score was done before treatment as a baseline; and 4 weeks after treatment.
  It was performed using the mean Karnofsky performance score

SECONDARY OUTCOMES:
Arterial blood gases evaluation | Arterial blood gases was done before treatment as a baseline; and 4 weeks after treatment.
  It included; Mean So2 (mm Hg), Mean PaO2 (mmHg), Mean PaCo2 (mm Hg).
Six minute walk distance test | Six minute walk test was done before treatment as a baseline; and 4 weeks after treatment.
  Six minute walk distance test was measured in minutes

IPD SHARING:
Plan to Share IPD: Undecided